CLINICAL TRIAL: NCT03833739
Title: A Prospective Randomized Clinical Trial to Compare Between Two Leveling and Alignment Protocols for the Treatment of Class II Division 2 Malocclusion
Brief Title: Comparison Between 2 Protocols for the Treatment of Class II Division 2 Malocclusion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jordan University of Science and Technology (Other)
Responsible Party: Principal Investigator, Mahmoud abuaysheh, Principal Investigator - Master student, Jordan University of Science and Technology
Allocation: Randomized | Model: Parallel | Purpose: Treatment
Other Study IDs: 461/2017
Record Dates: First submitted 2019-02-06; First posted 2019-02-07 (Actual); Last update posted 2019-02-21 (Actual); Status verified 2019-02

CONDITIONS: Class II Div 2 Incisal Relationship
Keywords: Class II division 2; Alignment; Leveling
MeSH Terms: conditions — Malocclusion, Angle Class II | interventions — Orthodontic Appliances, Fixed

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Upper Arch Treatment First (Experimental): Intervention : using fixed orthodontic pre-adjusted edgewise appliance in the upper and lower arches.
  starting treatment in the upper arch The upper ach was bonded for 28 patients and teeth alignment was started using round 0.014"NiTi arch wire. The 0.014"NiTi arch wire was placed into the slots of the brackets and tied with elastomers by figure of 8. Orthodontic treatment was continued in the upper arch with arch wire sequence of 0.014"NiTi, 0.018"NiTi, 0.016"X0.022"NiTi, 0.019"X0.025"NiTi, and 0.019"X0.025"stainless steel arch wires. The patients were followed up on a monthly basis until sufficient proclination of the upper incisors achieved to establish an overjet of at least 4 mm. After reaching the full working arch wire in lower arch (0.019" X 0.025"stainless steel wire), lateral cephalogram and study models were taken.
  Interventions: Device: Fixed appliance
- Lower Arch Treatment First (Experimental): Intervention : using fixed orthodontic pre-adjusted edgewise appliance in the lower arch and anterior bite plate in the upper arch.
  The lower arch was bonded after taking the pretreatment records. At the same appointment an anterior bite plate in the upper arch was delivered to prevent shearing off the mandibular incisor brackets and help in correction of anterior deep bite .After lower arch alignment and leveling in the same arch wire sequence as the other group and 0.019" X 0.025"stainless steel arch wire was reached, the anterior bite plate was removed and the upper arch was bonded. The same arch wire sequence was used in the upper arch as was used in the lower arch. When the full working arch wire (0.019" X 0.025"stainless steel arch wire) was reached in the upper arch, study models and lateral cephalogram were taken.
  Interventions: Device: Fixed appliance

INTERVENTIONS:
Device: Fixed appliance

SUMMARY:
The aim of this prospective study was to compare between two different treatment modalities of class II division 2; to start treatment in upper arch first until adequate overjet is obtained or to start in the lower arch first with removable anterior bite plane in upper arch.

DETAILED DESCRIPTION:
Fifty four subjects with class II division 2 participated in this study. The subjects were randomly divided into two groups; Group one (28 patients): orthodontic treatment with upper arch bond up first and lower arch was bonded when 4 mm overjet was reached. The treatment continued until 0.019 x 0.025 " stainless steel wires were reached in both arches. Group 2 (26 patients): orthodontic treatment with lower arch bond up first with removable anterior bite plane in upper arch. When 0.019 x 0.025" stainless steel wire was reached, the upper arch was bonded. The treatment continued until 0.019 x 0.025" stainless steel wires were reached. Three cephalograms were taken for each patient in both groups; pretreatment (T0) , after bonding the other arch (T1) and at the end of leveling and alignment in both arches (T2). Cephalometric measurements and superimpositions were made. Skeletal and dentoalveolar treatment changes were compared within and between the 2 groups.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 17 years and ≤ 26 years
* Class II division 2 malocclusion.
* Overjet (OJ) < 4 mm.
* Overbite (OB) covering more than half of the lower incisor height.
* Mild to moderate crowding with tooth contact displacement no more than 2 mm.
* Good oral hygiene and healthy periodontium.

Exclusion Criteria:-

* Systemic health problems and medications were taken.
* History of previous orthodontic treatment.

Ages: 17 Years to 26 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 54 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2018-01-01 (Actual); Study Completion 2018-11-01 (Actual)

PRIMARY OUTCOMES:
Upper and lower incisors proclination | 2 years
  Cephalometric analysis. Treatment changes in the values for upper and lower incisors in degrees, Upper incisor /Maxillary plane in degrees and lower incisors/Mandibular plane in degrees.

SECONDARY OUTCOMES:
Duration of treatment | 2 years
  Measurements of time of treatment in months
Pain perception | 2 years
  Using visual analogue scale. From 0 where is no pain to 10 with severe pain

CONTACTS AND LOCATIONS:
Overall Officials: Susan AlKhateeb, PhD, Principal Investigator — Jordan University of Science and Technology
Locations (1):
- Jordan University of Science and Technology Dental Teaching Clinics, Irbid, Jordan

IPD SHARING:
Plan to Share IPD: Undecided